CLINICAL TRIAL: NCT04441346
Title: Frequency and Risk Factors of Congestive Heart Failure in Dialysis Patients Attending Assiut University Hosptial
Brief Title: Frequency and Risk Factors of Congestive Heart Failure in Dialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Galal, Resident Doctor, internal medicine department, principal investigator, Assiut University
Other Study IDs: CHF in Dialysis patients
Record Dates: First submitted 2020-06-06; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients with recent hemodialysis(less than 6 month
  Interventions: Radiation: Echocardiography
- patients on hemodialysis more than 6 months and l
  Interventions: Radiation: Echocardiography
- patients on hemodialysis more than 5 years
  Interventions: Radiation: Echocardiography

INTERVENTIONS:
Radiation: Echocardiography — test that uses high frequency sound waves (ultrasound) to make pictures of your heart.

SUMMARY:
This study aims :

To assess the frequency of heart failure in patients with end-stage renal disease on regular dialysis.

To identify the risk factors of heart failure in patients with end-stage renal disease.

To assess the impact of duration of dialysis on heart failure and its prognosis

DETAILED DESCRIPTION:
Heart Failure is defined as a complex clinical syndrome that can result from any structural or functional cardiac disorder that impairs the ability of the ventricle to fill or eject blood with diagnosis relying on clinical examination and associated with significant mortality and morbidity. Congestive heart failure (CHF) is a cardiovascular complication in which the heart becomes unable to supply a sufficient amount of blood to meet the metabolic requirements and fulfill the body's oxygen demand.

CHF is an independent risk factor for early mortality in ESRD patients. More than half of all deaths among ESRD patients are due to cardiovascular disease (CVD). Cardiovascular changes secondary to renal dysfunction, including fluid overload, uremic cardiomyopathy, secondary hyperparathyroidism, anemia, altered lipid metabolism, and accumulation of gut microbiota-derived uremic toxins like trimethylamine N-oxidase (TMAO), contribute to the high risk for CVD in the ESRD population. Also, conventional hemodialysis (HD) itself poses myocardial stress and injury to the already compromised cardiovascular system in uremic patients.

The characteristics of cardiovascular dysfunction observed in dialysis patients are distinct from those noted in the general population. Although traditional cardiovascular risk factors in patients with end-stage renal disease (ESRD) are highly prevalent, they play only a partial role in the excessive cardiovascular morbidity and mortality of this population. The paradoxical association between several traditional risk factors, such as body mass index, blood pressure (BP) and serum cholesterol, and mortality have been previously reported.

In the ESRD population, Hemodialysis (HD) contributes itself to the development of CHF with sustained fluid overload a major cause of hypertension, heart failure, and mortality in patients with ESRD. We postulate that repeated myocardial micro-injury during maintenance hemodialysis may lead to irreversible cardiac dysfunction and subsequent heart failure and death in some patients.

ELIGIBILITY:
Inclusion Criteria:

* ESRD patient on regular hemodialysis

Exclusion Criteria:

* AKI patients on HD
* Patients discontinued therapy during the study period will be excluded.
* Patients with structural heart disease (congenital or valvular heart disease)
* Patients with obstructive or restrictive lung diseases.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Dialysis unit of Internal Medicine Department in Assiut University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 289 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
risk factors of CHF in hemodialysis patients | July 2020 to July 2021
  identification of risk factors using demographic and disease characteristics of the patient as age, gender, systolic and diastolic blood pressure, dialysis access, frequency and duration of HD
incidence of CHF in hemodialysis patients | July 2020 to July 2021
  identification of CHF in ESRD patients using echocardiography

SECONDARY OUTCOMES:
impact of duration of dialysis on heart failure | July 2020 to July 2021
  determine the extent of CHF in relation to duration of dialysis